CLINICAL TRIAL: NCT04524845
Title: Study of Biomechanical Parameters of Unloading Braces Used in the Treatment of Knee Osteoarthritis (BIOoSE)
Acronym: BIOoSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Collaborators: University Hospital of Saint-Etienne (Other); Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC25; 2017-A01963-50 (Other: ANSM)
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over, open labelled, monocentric, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rebel Reliever (Experimental): Rebel Reliever (RR) (Thuasne, Levallois Perret, France) with bilateral rigid frames and two hinges. The valgus correction was set by adjusting the medial and lateral frame lengths to a difference of two or three points as dictated by the participant's feeling and comfort. Six straps maintained the brace in place
  Interventions: Device: Rebel Reliever (RR)
- Action Reliever (Experimental): Action Reliever (AR) (Thuasne, Levallois Perret, France) made mainly from textile. Upper and lower straps were adjusted to the participant's feeling and comfort.
  Interventions: Device: Action Reliever
- Unloader One (Active Comparator): Unloader One (UO) (Össur, Reykjavik, Iceland), with unilateral frame and one hinge. Upper and lower straps were adjusted to the setting recommended by the fitting instructions and confirmed by the participant's sensation.
  Interventions: Device: Unloading brace
- No orthosis (No Intervention): Control condition without brace

INTERVENTIONS:
Device: Unloading brace — Participants underwent one session of gait analysis. The experimental protocol was divided in four conditions, the control condition without brace (NO), and then three conditions with the different braces tested in a randomized order.
  For each condition, the participant was fitted with the brace by the same experimenter and equipped with 19/20 retro-reflective markers (without/with brace) on the pelvis and the investigated leg for motion analysis. After a short recording in a fixed standing position (static trial), each participant carried out at least three barefoot walking trials of a few meters long at a self-selected pace. The walking trial was validated if a complete gait cycle occurred on the two 90cm x 90 cm force plates recording the ground reaction forces. After each condition, the participant had to assess knee pain.
  Arms: Unloader One
Device: Rebel Reliever (RR) — Rebel Reliever (RR) (Thuasne, Levallois Perret, France)
  Arms: Rebel Reliever
Device: Action Reliever — Action Reliever (AR) (Thuasne, Levallois Perret, France)
  Arms: Action Reliever

SUMMARY:
Osteoarthritis is a chronic disease affecting millions of people worldwide, and knee is the second most affected site. Knee osteoarthritis is characterized by knee pain, loss of motion, disability, and muscle weakness, all factors contributing to gait alterations, and impacting greatly the patients quality of life. In the absence of curative treatment, pharmacological and non-pharmacological symptomatic treatments are prescribed to maintain this QoL, and therefore delay surgery to more appropriate window of opportunity later in life.

The aim of the study was to investigate the acute effects of three braces, using different unloading strategies, on gait kinematic and kinetic parameters, as well as pain in patients with medial knee ostoeoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* unilateral medial KOA classified II or III on the Kellgren-Lawrence scale
* varus misalignment with a joint space of at least two finger breadths
* pain level equal or higher than 30 mm on a 100 mm visual analog scale
* informed written consent

Exclusion Criteria:

* limited ability to walk
* normoaxial knee alignment
* intra-articular injection of a local treatment including corticosteroids in the 3 months or hyaluronic acid in the 6 months preceding its inclusion or analgesic or NSAID treatment with a wash-out period equal to 5 half-lives of the drug concerned
* undergoing physiotherapy
* cognitive disorders or behavioral disorders (opposition, agitation, dementia)
* arteriopathy of the lower limbs
* skin disorders contraindicating the wearing of rigid orthotics
* severe varicosity preventing the regular wearing of unloading brace

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Knee Adduction Moment | Day : 1
  Main parameter determined from the force platforms:
  - Position of the center of gravity
  By coupling the techniques of kinematic measurement and ground reaction force, we obtain the Moment of Adduction (or KAM) when walking
Knee Adduction Moment | Day : 1
  Main parameter determined from the force platforms:
  - Impact force and vertical propulsive force. By coupling the techniques of kinematic measurement and ground reaction force, we obtain the Moment of Adduction (or KAM) when walking

SECONDARY OUTCOMES:
Perceived pain | Day: 1
  The pain is self-assessed by the patient using a visual analogue scale graduated from 0 to 10: the analogue scale is presented to the patients, who will mark the level of pain felt during the works under each of the study conditions.
Adduction/abduction angles | Day: 1
  Adduction/abduction angles (in particular A1 and A2, corresponding to the two vertical GRF maxima, as well as the adduction angle during standing (A0)), were measured (deg) under each condition.
Impact and propulsive reaction force of the ground | Day: 1
  The impact force and the propulsive reaction force of the ground (N / kg) were measured during walking under each condition. F1 corresponds to the load response peak and F2 to the terminal stance peak during gait,
Step length | Day: 1
  The length of the step (m) was measured during walking under each condition.
Walking speed | Day: 1
  The walking distance (km/h) was measured during walking under each condition.
Satisfaction related to the device | Day: 1
  A satisfaction survey is filled by the patient in order to assess the positioning of unloading brace, comfort, esthetic and global satisfaction of devices

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Thomas, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Saint-Etienne Jean Monnet University, Saint-Etienne, France